CLINICAL TRIAL: NCT00057720
Title: Phase 3 Randomized Study of TLK286 (Telcyta) Versus Doxil/Caelyx or Hycamtin as Third-Line Therapy in Platinum Refractory or Resistant Ovarian Cancer [ASSIST-1 (Assessment of Survival In Solid Tumors-1)]
Brief Title: TLK286 (Telcyta) vs. Doxil/Caelyx or Hycamtin in Platinum Refractory or Resistant Ovarian Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Telik (Industry)
Responsible Party: Gail Brown, MD Chief Medical Officer, Telik, Inc
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: TLK286.3017; NCT00078884 (obsolete NCT alias)
Record Dates: First submitted 2003-04-07; First posted 2003-04-08 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2006-05

CONDITIONS: Ovarian Neoplasms
Keywords: ovary
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Injections; Topotecan

INTERVENTIONS:
Drug: TLK286 HCl for injection
Drug: topotecan hydrochloride for injection
Drug: doxorubicin HCl liposome injection

SUMMARY:
The purpose of this study is to demonstrate superiority in survival in favor of TLK286 as compared to active control therapy with Doxil/Caelyx or Hycamtin in the intent-to-treat (ITT) populations.

ELIGIBILITY:
Inclusion criteria include:

* Considered platinum refractory or resistant according to standard criteria
* Progressed during or following completion of one second-line treatment with Doxil/Caelyx or Hycamtin
* Histologically or cytologically confirmed diagnosis of epithelial cancer of the ovary, fallopian tube, or primary peritoneal cancer
* Measurable disease according to RECIST criteria with documented tumor progression

Exclusion criteria include:

* Treatment with second-line chemotherapy other than Doxil/Caelyx or Hycamtin
* History of whole pelvis radiation therapy within 12 months of enrollment
* Clinically significant cardiac disease
* Evidence of gross hematuria at the time of study entry
* Any signs of intestinal obstruction interfering with nutrition at the time of study entry
* Pregnant or lactating women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440
Dates: Start 2003-06; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (311):
- United States (225):
  - Little Rock Hematology Oncology Associates, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Baldwin Park, California
  - Providence Saint Joseph Medical Center, Burbank, California
  - Marilyn Norton, M. D., Chula Vista, California
  - Rosalba Rodriguez, M. D., Chula Vista, California
  - Bay Area Research Cancer Group, Concord, California
  - Southwest Cancer Care, Escondido, California
  - California Oncology of the Central Valley, Fresno, California
  - Kaiser Permanente Oncology Clinical Trials Program, Hayward, California
  - Gynecologic Oncology Associates, La Jolla, California
  - Grossmont Hospital, La Mesa, California
  - Sharp Rees-Stealy, La Mesa, California
  - LLU Faculty Medical Offices, Loma Linda, California
  - LLU Faculty Meidical Offices, Loma Linda, California
  - Loma Linda University Medical Center, Loma Linda, California
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Women's Cancer Center - Community Hospital Los Gatos, Los Gatos, California
  - Southwest Cancer Care, Murrieta, California
  - Gyncologic Oncology Associates, Newport Beach, California
  - Kaiser Permanente Oncology Clinical Trials Program, Oakland, California
  - N. County Oncology Medical, Oceanside, California
  - Southwest Cancer Care, Poway, California
  - Kaiser Permanente Oncology Clinical Trials Program, Redwood City, California
  - Kaiser Permanente Oncology Clinical Trials Program, Roseville, California
  - Kaiser Permanente Oncology Clinical Trials Program, Sacramento, California
  - Southern California Permanente Medical Group, San Diego, California
  - Medical Oncology Associates-SD, San Diego, California
  - Sharp Healthcare Clinical Oncology Research, San Diego, California
  - Sharp Memorial Hospital, San Diego, California
  - Sharp Rees-Stealy, San Diego, California
  - Kaiser Permanente Oncology Clinical Trials Program, San Francisco, California
  - Kaiser Permanente Oncology Clinical Trials Program, San Rafael, California
  - Kaiser Permanente Oncology Clinical Trials Program, Santa Clara, California
  - Kaiser Permanente Oncology Clinical Trials Program, Santa Rosa, California
  - Kaiser Permanente Oncology Clinical Trails Program, Santa Teresa, California
  - Kaiser Permanente Oncology Clinical Trials Program, South San Francisco, California
  - Kaiser Permanente Oncology Clinical Trials Program, Vallejo, California
  - Kaiser Permanente Oncology Clinial Trials Program, Walnut Creek, California
  - Whittingham Cancer Center at Norwalk Hospital, Norwalk, Connecticut
  - Hematology Oncology, P.C., Stamford, Connecticut
  - The Center for Hematology-Oncology, Boca Raton, Florida
  - The Center for Hematology-Oncology, Delray Beach, Florida
  - Memorial Regional Hospital, Hollywood, Florida
  - Sheridan Clinical Research, Inc., Hollywood, Florida
  - University of Florida Health Science Center/Jacksonville, Jacksonville, Florida
  - Florida Hospital, Orlando, Florida
  - Gynecologic Oncology, Orlando, Florida
  - Florida Hospital Memorial Division, Cancer Care Center, Ormond Beach, Florida
  - Florida Hospital Memorial Division, Ormond Beach, Florida
  - Palm Beach Cancer Institute, Palm Beach Gardens, Florida
  - Gynecologic Oncology Associates, Pembroke Pines, Florida
  - Hematology/Oncology Associates of Treasure Coast, Port Saint Lucie, Florida
  - Women's Cancer Research Foundation, Inc., South Miami, Florida
  - Palm Beach Cancer Institute, Wellington, Florida
  - Palm Beach Cancer Institute, West Palm Beach, Florida
  - Suburban Hematology Oncology, Duluth, Georgia
  - Suburban Hematology-Oncology Associates, Lawrenceville, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Suburban Hematology Oncology, Snellville, Georgia
  - Kaiser Permanente - Moanalua Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - Univ. of Hawaii, Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - North Shore Oncology Hematology Associates, Barrington, Illinois
  - MacNeal Cancer Center, Berwyn, Illinois
  - Swedish Covenant Cancer Center, Chicago, Illinois
  - Hematology Oncology Associates of Illinois (HOAI), Chicago, Illinois
  - Cancer Care Specialists of Central IL, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Cancer Care Specialists of Central IL-Crossroads Cancer Care Center, Effingham, Illinois
  - Joliet Oncology-Hematology Associates, Ltd., Flossmoor, Illinois
  - Joliet Oncology-Hematology Associates, Ltd., Joliet, Illinois
  - North Shore Oncology Hematology Associates - Deerpath Medical Associates, Lake Forest, Illinois
  - North Shore Oncology Hematology Associates, Libertyville, Illinois
  - North Shore Oncology Hematology Associates, McHenry, Illinois
  - Joliet Oncology-Hematology Associates, Ltd., Morris, Illinois
  - Hematology Oncology Associates of Illinois (HOAI), Skokie, Illinois
  - Midwest Cancer Research Group, Inc., Skokie, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Michiana Hematology Oncology, Elkhart, Indiana
  - Indiana Cancer Pavilion, Indianapolis, Indiana
  - Indiana University Medical Center, Indianapolis, Indiana
  - St. Vincent Gynecologic Oncology, Indianapolis, Indiana
  - St. Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - St. Vincent Hospital and Helath Care Center, Indianapolis, Indiana
  - Michiana Hematology Oncology, South Bend, Indiana
  - St. Joseph's Regional, South Bend, Indiana
  - Saint Joseph's Regional, South Bend, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Iowa, Iowa City, Iowa
  - Research Support Personnel, LLC, Wichita, Kansas
  - Associates in Women's Health, Wichita, Kansas
  - Oncology/Hematology Care, Inc., Crestview, Kentucky
  - Univ. of Louisville, Div. of Gynecologic Oncology, Louisville, Kentucky
  - Hematology and Oncology Specialists, LLC, Covington, Louisiana
  - OncRx (Pharmacy), Metairie, Louisiana
  - Hematology and Oncology Specialists, LLC, New Orleans, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - LSU Health Sciences Center, Shreveport, Louisiana
  - Sinai Cancer Institute, Baltimore, Maryland
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - St. Elizabeth's Med. Ctr., Boston, Massachusetts
  - St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary's Duluth Clinic, Duluth, Minnesota
  - Ellis Fischel Cancer Center, Columbia, Missouri
  - St. Louis University, Dept. of Ob-Gyn and Women's Health, St Louis, Missouri
  - Gynecology & Oncology Consultants, PC, St Louis, Missouri
  - Saint John's Mercy Hospital, St Louis, Missouri
  - Deaconess Billings Clinic, Billings, Montana
  - Hematology & Oncology Centers Northern Rockies, Billings, Montana
  - Hematology Oncology Centers of the Northern Rockies, Butte, Montana
  - Horizon's West Medical Group, Scottsbluff, Nebraska
  - Nevada Cancer Center, Las Vegas, Nevada
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - The Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - UNM Cancer Research and Treatment Center, Albuquerque, New Mexico
  - Benjamin Schwartz, M.D., Babylon, New York
  - The Mary Imogene Bassett Hospital, Cooperstown, New York
  - Med-Onc/Hem, Malone, New York
  - Hematology-Oncology Associates of Rockland, New City, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - North Shore-Long Island Jewish Health System/Medical Center, New Hyde Park, New York
  - Bellevue Hospital Center, New York, New York
  - Comprehensive Cancer Center Medical Practice Offices, New York, New York
  - New York University Medical Center - Tisch Hospital, New York, New York
  - NYU School of Medicine, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - The Union State Bank Cancer Center at Nyack Hospital, Nyack, New York
  - Gynecologic-Oncology, Rochester, New York
  - Good Samaritan Hospital Medical Center, West Islip, New York
  - South Bay OB/GYN, West Islip, New York
  - Blumenthal Cancer Center, Charlotte, North Carolina
  - Presbyterian Gynecologic Oncology, Charlotte, North Carolina
  - Presbyterian Hospital Center for Cancer Research, Charlotte, North Carolina
  - Piedmont Hematology Oncology Assoc., PA-Salem Research Group, Winston-Salem, North Carolina
  - Salem Research Group, Inc., Winston-Salem, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Odyssey Research Services, Bismarck, North Dakota
  - Dakota Cancer Institute, Fargo, North Dakota
  - Odyssey Research Services, Fargo, North Dakota
  - Oncology/Hematology Care, Inc., Cincinnati, Ohio
  - Barrett Cancer Center, Cincinnati, Ohio
  - UC Physician's Medical Arts Bldg., Cincinnati, Ohio
  - UC Physician's Medical Arts Building, Cincinnati, Ohio
  - University Hospital, Cincinnati, Ohio
  - Metro Health Medical Center, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Mid-Ohio Oncology Hematology St. Anne's, Columbus, Ohio
  - Mid Ohio Oncology Hematology, Columbus, Ohio
  - Mid-Ohio Oncology Hematology, Columbus, Ohio
  - Gynecologic Oncology, Columbus, Ohio
  - Mount Carmel Health, Columbus, Ohio
  - Wright State Univ. School of Medicine, Dayton, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - OU Medical Center - Everett Tower, Oklahoma City, Oklahoma
  - OU Physicians' Bldg., Oklahoma City, Oklahoma
  - Presbyterian, Oklahoma City, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Kaiser Permanente Nw, Oncology Research, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Oregon Health Science University, Portland, Oregon
  - Abington Mem. Hospita/Rosenfield Cancer Center, Abington, Pennsylvania
  - Advanced Imaging, Dunmore, Pennsylvania
  - Hematology & Oncology Associates of NEPA, Dunmore, Pennsylvania
  - Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - Viewmont Medical Services, Scranton, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Mercy Health Partners, Scranton, Pennsylvania
  - Moses Taylor Hospital, Scranton, Pennsylvania
  - Associates in Hematology-Oncology, P.C., Upland, Pennsylvania
  - Carolina Center of Gynecologic Oncology, PA, Charleston, South Carolina
  - South Carolina Oncology Associates, PA, Columbia, South Carolina
  - Gynecologic Oncology Research and Development, Greenville, South Carolina
  - Gynecologic Oncology Research and Development, Spartanburg, South Carolina
  - Sioux Valley Clinic Clinical Research Center, Sioux Falls, South Dakota
  - Sioux Valley Clinic Oncology, Sioux Falls, South Dakota
  - Sioux Valley Hospital - North Center Radiology, Sioux Falls, South Dakota
  - Sioux Calley Clinic OBGYN Ltd., Sioux Falls, South Dakota
  - Chattanooga Oncology & Hematology Associates, P.C., Chattanooga, Tennessee
  - Memorial Hospital, Chattanooga, Tennessee
  - The Consultant Group, Franklin, Tennessee
  - The Sarah Cannon Cancer Center/Tennessee Oncology, PLLC, Gallatin, Tennessee
  - The Sarah Cannon Cancer Center/Tennessee Oncology, PLLC, Hermitage, Tennessee
  - Saint Mary's Health System, Inc., Knoxville, Tennessee
  - Hall and Martin, M.D.'s, P.C., Knoxville, Tennessee
  - Fort Sanders Parkwest Medical Center, Knoxville, Tennessee
  - The Sarah Cannon Cancer Center/Tennessee Oncology, PLLC, Lebanon, Tennessee
  - The Sarah Cannon Cancer Center/Tennessee Oncology, PLLC, Murfreesboro, Tennessee
  - The Sarah Cannon Cancer Center/Tennessee Oncology, PLLC, Nashville, Tennessee
  - The Consultant Group, Nashville, Tennessee
  - The Sarah Cannon Cancer Center/Tennessee Oncology, PLLC, Smyma, Tennessee
  - Amarillo Cancer Center, Amarillo, Texas
  - Arlington Cancer Center, Arlington, Texas
  - Dallas Oncology Consultants, Dallas, Texas
  - Texas Cancer Associates, Dallas, Texas
  - Texas Oncology, PA, Fort Worth, Texas
  - Southwest Fort Worth Cancer Center, Fort Worth, Texas
  - Univ. of TX, MD Anderson Cancer Center, Houston, Texas
  - Danville Hematology and Oncology, Inc., Danville, Virginia
  - Western Washington Oncology, Aberdeen, Washington
  - Western Washington Oncology, Centralia, Washington
  - Covington Multicare - Oncology Clinic, Covington, Washington
  - Western Washington Oncology, Olympia, Washington
  - Western Washington Oncology, Shelton, Washington
  - Allenmore Hospital - Hematology Oncology Clinic, Tacoma, Washington
  - MultiCare Health System - Medical Oncology, Tacoma, Washington
  - Chippewa Falls Cancer Center, Chippewa Falls, Wisconsin
  - Regional Cancer Center, Eau Claire, Wisconsin
  - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
  - Saint Joseph's Hospital, Marshfield, Wisconsin
  - Wisconsin Rapid Cancer Center, Marshfield, Wisconsin
  - Merrill Cancer Center, Merrill, Wisconsin
  - Medical Consultants, Ltd., Milwaukee, Wisconsin
  - Marshfield Clinc - Lakeland Center, Minocqua, Wisconsin
  - Marshfield Clinic - Lakeland Center, Minocqua, Wisconsin
  - Diagnostic Radiology Associates, Rice Lake, Wisconsin
  - Lakeview Medical Center, Rice Lake, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - Saint Michael Hospital, Stevens Point, Wisconsin
  - Wausau Cancer Center, Wausau, Wisconsin
  - Hematology Oncology Centers of the Northern Rockies, Cody, Wyoming
  - Hematology Oncology of the Northern Rockies, Sheridan, Wyoming
- Argentina (13):
  - Hospital Italiano Regional del Sur, Bahía Blanca, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires, Buenos Aires
  - Sanatorio Municipal Dr. Julio Mendez, Buenos Aires, Buenos Aires
  - Hospital General de Agudos "Carlos G. Durand", Buenos Aires, Buenos Aires
  - Complejo Medico de la Policia Federal Argentina "Churruca-Visca", Buenos Aires, Buenos Aires
  - Hospital de Oncologia Maria Curie, Buenos Aires, Buenos Aires
  - Policlinica Privada Instituto de Medicina Nuclear, Buenos Aires, Buenos Aires
  - Hospital General de Agudos Donacion F. Santojanni, Capital Federal, Buenos Aires
  - Hospital Universitario Austral, Pilar, Buenos Aires
  - ISIS Clinica Especializada, Santa Fe, Santa Fe Province
  - Hospital Donacion Francisco Santojanni, Buenos Aires
  - Complejo Medico de la Policia Federal Argentina "Churruca-Visca", Buenos Aires
  - Sociedad de Beneficencia Hospital Italiano, Córdoba
- Belgium (7):
  - Algemeen Ziekenhuis Antwerpen, Lindedreef, Antwerpen
  - Universitaire Ziekenhuis Antwerpen, Wilrijkstraat, Edegem
  - University Hospital Gasthuisberg, Herestraat, Leuven
  - AZ-VUB Dienst Oncologie, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Gent., Ghent
  - Centre Hospitalier Regional de la Citadelle, Liège
- Brazil (12):
  - Instituto do Cancer do Ceara, Fortaleza, Ceará
  - Hospital Vera Cruz, Belo Horizonte, Minas Gerais
  - Hospital Luxemburgo, Belo Horizonte, Minas Gerais
  - Hospital de Clinicas da Universidade Federal do Parana, Curitiba, Paraná
  - Centro de Tratamento Oncologico de Londrina, Londrina, Paraná
  - Hospital de Clinicas de Porto Alegre, Bairro Bom Fim, Porto Alegre
  - INCA Hospital de Oncologia Clinica, Rio de Janeiro, Rio de Janeiro
  - Instituto Arnaldo Vieira de Carvalho, São Paulo, São Paulo
  - Hospital do Cancer - A.C. Camargo, São Paulo, São Paulo
  - Unifesp/Epm, São Paulo, São Paulo
  - Hospital das Clinicas de Sao Paulo-FMUSP, São Paulo, São Paulo
  - Instituto de Saude e Bem Estar da Mulher, São Paulo, São Paulo
- Chile (2):
  - Clinica Santa Maria, Santiago, Santiago de Chile
  - Servicio de Oncologia-Hospital Clinico Unversidad de Chile, Independencia, Santiago Metropolitan
- Czechia (8):
  - Fakultni nemocnice Olomouc, Onkologicka klinika, Pardubice, Olomouc
  - Krajska nemocnice Pardubice, Oddeleni radiacni onklogie, Kyjevska 44, Pardubice
  - Fakultni Nemocnice - Onkologicka Klinika, Doudlevecka 69, Plzen
  - Vseobecna Fakultni Nemocnice - Onkologicka Klinika, Unemocnice, Prague
  - Batova krajska nemocnice Zlin, prispevkova organizace, Onkologicke oddeleni, Havlickovo Nabrezi 600, Zlín
  - Batova krajska nemocnice Zlin, prispevkova organizace, Radiodiagnosticke oddeleni, Havlickovo Nabrezi, Zlín
  - Masarykuv Onkologicky Ustav, Brno
  - Fakultni nemocnice, Onkologicka klinika, Pilsen
- Germany (8):
  - Universitatsklinikum Charite - Campus Virchow-Klinikum, Berlin
  - St. Vincentius Kliniken, Karlsruhe
  - St. Vincentius Kliniken - Frauenkinik, Karlsruhe
  - St. Vincentius Kliniken - Radiology, Karlsruhe
  - Klinikum GroBhadern-Institut fur Radiologie, Munich
  - Klinikum GroBhadern-Zentrum fur Frauenheilkunde, Munich
  - Universitaets-Frauenklinik Ulm, Ulm
  - Dr. Horst-Schmidt-Kliniken GmbH, Wiesbaden
- Hungary (7):
  - Semmelweis University, 1st Dept. of Obstetrics and Gynaecology, Baross
  - Uzsoki Street Hospital Dept. of Radiooncology, Budapest
  - Faculty of Gynaecologycal Oncology/Univ. of Debrecen, Debrecen
  - Baranya County Hospital, Pécs
  - Baranya County Hospital - Department of Oncology, Rakoczi
  - Baranya County Hospital - Department of Radiology, Rakoczi
  - SZTE, Department of Oncotherapy, Szeged
- Oncology Dept., University Floor, Belfast City Hospital, Belfast, Ireland
- Netherlands (2):
  - Vrije Universiteit Medical Centre (VUMC), HV Amsterdam
  - University Medical Centre Nijmegen (UMCN), Nijmegen
- South Africa (6):
  - Panorama Medical Centre, Panorama, Cape Town
  - Hopelands Cancer Centre, Overport, Durban
  - Medical and Dental Centre, Rosebank, Johannesburg
  - Rosebank Oncology Centre, Saxonwold, Johannesburg
  - Wilgers Oncology Centre, Die Wilgers X14, Pretoria
  - Eastern Cape Oncology Research Centre, Port Elizabeth
- Spain (8):
  - Servicio Oncologia Hospital General Vall d'HebronPaseo, Vall d'Hebron, Barcelona
  - Instituto Valenciano de Oncologia (IVO), Profesor Beltran Baguena, Valencia
  - Hospital Clinic i Provincial de Barcelona - Servicio de Oncologia Medica, Barcelona
  - Hospital Clinic i Provincial, Barcelona
  - Hospital General de Guadalajara, Guadalajara
  - Servicio de Oncologia, Madrid
  - Instituto Valenciano de Oncologia (IVO) Servicio de Oncologia, Valencia
  - Instituto Valenciano de Oncologia (IVO) Servicio de Radiologia, Valencia
- United Kingdom (12):
  - Department of Cancer Medicine - Ninewells Hospital & Medical School, Scotland, Dundee
  - Dept. of Med. Oncology/The Royal Marsden Hospital, Sutton, Surrey
  - St. Chad's Outpatients Unit, City Hospital, Birmingham
  - United Bristol Healthcare Trust - Bristol Oncology Centre, Bristol
  - Beatson Oncology Centre, Glasgow
  - Beatson Oncology Unit, Glasgow
  - Medical Oncology - Guy's and St. Thomas' Hospital, London
  - Department of Medicine-Royal Marsden Hospital, London
  - Department of Medical Oncology, Christie Hospital, Manchester
  - Medical Oncology (NCCT) - Newcastle General Hospital, Newcastle upon Tyne
  - Dorset Cancer Centre - Poole Hospital, Poole
  - Velindre NHS Trust - Velindre Hospital, Wales